CLINICAL TRIAL: NCT02655640
Title: The Impact of Illness Perceptions and Their Determinants on Health Related Outcomes in Patients With Systemic Lupus Erythematosus and Systemic Sclerosis
Brief Title: The Impact of Illness Perceptions on Health Related Outcomes in Patients With Lupus and Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S58458
Record Dates: First submitted 2015-12-01; First posted 2016-01-14 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2015-09

CONDITIONS: Lupus Erythematosus, Systemic; Scleroderma, Systemic
Keywords: illness perceptions
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lupus: Characteristics of patients with Systemic Lupus Erythematosus. No interventions will be administered. Patients will be asked to complete questionnaires.
  Interventions: Other: Questionnaires
- Scleroderma: Characteristics of patients with Systemic Sclerosis. No interventions will be administered. Patients will be asked to complete questionnaires.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires will be provided to patients

SUMMARY:
This research project has the overall objective to investigate the direction of the associations between illness perceptions, their influencing factors and health-related outcomes. Moreover, the investigators want to look at the direction of the associations between illness perceptions and health related outcomes such as psychological and physical functioning in patients with Systemic Lupus Erythematosus (SLE) and Systemic Sclerosis (SSc). The investigators want to know whether the outcome variables anxiety, depression, physical (dis) functioning are influenced by illness perceptions or vice versa. Not only the patients' illness perceptions but also the illness perceptions of the General Practitioners (GP) and rheumatologists will be investigated. The researchers want to know if the doctors' perceptions have an impact on the physical and psychological functioning of the patient or vice versa. Much research in the field of illness perceptions is cross-sectional in nature which means that the direction of the relationships between variables is not known.

DETAILED DESCRIPTION:
This is a single center academic study at two timepoints with an interval of 12 months. The data collection includes demographic variables, patient-reported variables, clinical variables and healthcare professionals-reported variables. All SSc and SLE patients who meet the inclusion criteria and are monitored by the rheumatology consultation in the University Hospitals Leuven will be contacted to participate in the study. Patients will be informed of the purpose of the study and what is expected of them. If they agree to participate they will also be asked to sign the Informed Consent form to send together with the completed questionnaire by mail.

After the patient gives his/her agreement to participate his/ her GP and rheumatologist will be asked to fill out the Revised Illness Perception Questionnaire for Healthcare Professionals (IPQ-R HP). This is a questionnaire that measures the perception of the doctor about the disease condition of their patient.

Data will be collected and kept by the investigator for analysis after complete coding. The obtained data will be analyzed using statistical methods.

With this study the investigators want to give an answer on 4 research questions:

1. Are there differences in perceptions between GP's and rheumatologists?
2. What is the direction of the associations between the illness perceptions of the physicians and patients?
3. What is the direction of the associations between the illness perceptions of a patient with SLE or SSc and psychological and physical functioning?
4. What is the direction of the associations between the illness perceptions of the physician and the psychological and physical functioning of the patient?

ELIGIBILITY:
Inclusion Criteria:

* Before participation the patient gives informed consent.
* The medical condition of the patient allows him/her to complete a questionnaire
* The patient does not have a severe psychiatric comorbidity
* The patient can complete questionnaires in Dutch

Exclusion Criteria:

* no exclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Firstly a list will be created of all patients with lupus and systemic sclerosis who are in follow-up at the reumatology department in UZ Leuven. Afterwards all patients who fulfill the inclusion criteria will be selected. The patients who are included will be informed by mail and they will be asked to participate. When they agree for participating then they will be asked to complete an informed consent form.
  Hereafter the general practitioner and rheumatologist will be contacted to complete the IPQ-R HP (an illness perception questionnaire for Healthcare professionals)
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Anxiety | 12 months
  Anxiety will be measured with the Hospital Anxiety and Depression Scale.
Depression | 12 months
  Depression will be measured with the Hospital Anxiety and Depression Scale.
General Health Status | 12 months
  General Health Status will be measured with the EuroQol 5 dimensions.

SECONDARY OUTCOMES:
Illness perceptions of the general practitioner of a particular patient with SLE or SSc | 12 months
  This will be measured with the IPQ-R HP (revised Illness Perception Questionnaire for Healthcare Professionals)
Illness perceptions of the rheumatologist of a particular patient with SLE or SSc | 12 months
  This will be measured with the IPQ-R HP (revised Illness Perception Questionnaire for Healthcare Professionals)

CONTACTS AND LOCATIONS:
Overall Officials: Rene Westhovens, MD, PhD, Principal Investigator — UZ Leuven

REFERENCES:
- [Background] Petrie KJ, Jago LA, Devcich DA. The role of illness perceptions in patients with medical conditions. Curr Opin Psychiatry. 2007 Mar;20(2):163-7. doi: 10.1097/YCO.0b013e328014a871. PMID 17278916
- [Background] 2. Broadbent E. Illness perceptions and health: innovations and clinical applications. Soc Personal Psychol Compass 2010, 4(4):256-266.
- [Background] Leventhal, H, Meyer D, Nerenz D. The common-sense representation of illness danger. In S. Rachman (Ed.), Medical psychology 1980, Vol. 2: pp. 7-30. New York: Pergamon.
- [Background] Lau RR, Bernard TM, Hartman KA. Further explorations of common-sense representations of common illnesses. Health Psychol. 1989;8(2):195-219. doi: 10.1037//0278-6133.8.2.195. PMID 2737174
- [Background] Moss-Morris R, Weinman J, Petrie KJ, Horne R, Cameron LD, Buick D. The Revised Illness Perception Questionnaire (IPQ-R). Psychol Health 2002, 17(1):1-16.
- [Background] Benyamini, Y. Health and illness perceptions. In H. Friedman (Ed.), The oxford handbook of health psychology 2011, pp. 281-314. New York: Oxford University Press.
- [Background] Petrie KJ, Weinman J. Patients' perception of their illness: the dynamo of volition in health care. Curr Dir Psychol Sci 2012, 21(1):60-65
- [Background] Arat S, Verschueren P, De Langhe E, Smith V, Vanthuyne M, Diya L, Van den Heede K, Blockmans D, De Keyser F, Houssiau FA, Westhovens R. The association of illness perceptions with physical and mental health in systemic sclerosis patients: an exploratory study. Musculoskeletal Care. 2012 Mar;10(1):18-28. doi: 10.1002/msc.223. Epub 2011 Nov 11. PMID 22076953
- [Background] Daleboudt GM, Broadbent E, McQueen F, Kaptein AA. Intentional and unintentional treatment nonadherence in patients with systemic lupus erythematosus. Arthritis Care Res (Hoboken). 2011 Mar;63(3):342-50. doi: 10.1002/acr.20411. Epub 2010 Nov 30. PMID 21120967
- [Background] Daleboudt GM, Broadbent E, McQueen F, Kaptein AA. The impact of illness perceptions on sexual functioning in patients with systemic lupus erythematosus. J Psychosom Res. 2013 Mar;74(3):260-4. doi: 10.1016/j.jpsychores.2012.11.004. Epub 2012 Nov 21. PMID 23438719
- [Derived] Arat S, Rassart J, Moons P, Luyckx K, Vandenberghe J, Westhovens R. Prospective associations between illness perceptions and health outcomes in patients with systemic sclerosis and systemic lupus erythematosus: a cross-lagged analysis. Rheumatol Adv Pract. 2018 Mar 6;2(1):rky007. doi: 10.1093/rap/rky007. eCollection 2018. PMID 31431956
- [Derived] Arat S, Lenaerts JL, De Langhe E, Verschueren P, Moons P, Vandenberghe J, Taelman V, Westhovens R. Illness representations of systemic lupus erythematosus and systemic sclerosis: a comparison of patients, their rheumatologists and their general practitioners. Lupus Sci Med. 2017 Nov 14;4(1):e000232. doi: 10.1136/lupus-2017-000232. eCollection 2017. PMID 29177061